CLINICAL TRIAL: NCT06603116
Title: Evaluation of the Clinical Performance of Bioactive Giomer Restoration in Class II Cavities After One Year and in Vitro Investigation of the Surface Roughness
Brief Title: Evaluation of the Clinical Performance of Bioactive Giomer Restoration in Class II Cavities After One Year
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Noha Taher, Assistant lecturer at operative department, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTaher
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dental Restoration Failure
Keywords: Bioactive Giomer restoration; Nano hybrid composite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bioactive Giomer restoration. (Experimental): material applied according to manufacturer instructions. BEAUTIFIL II LS applied directly into the cavity and create the shape desired in layers not exceeding 2 mm and light cured for 20 seconds
  Interventions: Other: treatment of class two cavities
- Nano-hybrid Composite restoration. (Active Comparator): applied to the cavity use the conventional incremental technique according to manufacturer instruction
  Interventions: Other: treatment of class two cavities

INTERVENTIONS:
Other: treatment of class two cavities — restorations in class 2 cavities

SUMMARY:
Assess the clinical performance of the bioactive Giomer restoration in class II cavities after one year using FDI criteria for assessment of dental restorations. Moreover, the surface roughness will be investigated in-vitro using profilometer

DETAILED DESCRIPTION:
* Patients will be selected according to the following inclusion and exclusion criteria from the outpatient Operative clinic, Faculty of Dental Medicine for Girls, Al-Azhar University.
* The patients will be informed about the purpose of the investigation, the clinical procedures and the advantages/risks of the applied materials and techniques. A written informed consent form will be signed from patients prior to study initiation.
* Co-operative patients of age range 20-30 years old with no gender prediction, The patients will be divided into two groups Group (1): Bioactive Giomer restoration. Group (2): Nano-hybrid Composite restoration. Restoration will be evaluated using FDI criteria (functional and biological properties) All the restorations will be clinically evaluated after 1 week (baseline),3 month, 6 months,12 months.

data collected and statistically analyzed

ELIGIBILITY:
Inclusion Criteria:

* • Each patient should have at least two proximal carious lesions on both sides in the posterior teeth.

  * Adjacent and opposing natural teeth should be present.
  * Patient should be willing to return for follow-up examination and evaluation.

Exclusion Criteria:

* • Patient with poor oral hygiene and motivation.

  * Patient with unrealistic expectations.
  * Patients with disabilities, systemic diseases or severe medically compromised, bruxism, clenching or temporomandibular joint disorders and patients with allergy to any components of the materials.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
evaluation of restorations of class two cavities | from one week to one year
  Measured used FDI criteria

CONTACTS AND LOCATIONS:
Overall Officials: Maha Niazy, PHD, Study Director — Faculty of Dental Medicine for Girls, Al-Azhar University, Egypt
Locations (1):
- Faculty of Dental Medicine for Girls, Al-Azhar University, Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No